CLINICAL TRIAL: NCT06366971
Title: The Effect of Pelvic Proprioceptive Neuromuscular Facilitation Techniques in Patients With Sacroiliac Joint Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Hikmet Ucgun, Assistant Professor, Atlas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: auhucgun01
Record Dates: First submitted 2024-04-05; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Sacroiliac Joint Dysfunction
Keywords: flexibility; mobility; pain; proprioceptive neuromuscular facilitation; sacroiliac joint dysfunction
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group will receive exercise training consisting of pelvic PNF techniques in addition to patient education which consisting of basic lumbar stabilization exercises 3 days a week for 6-weeks.
  Interventions: Other: The Patient Education; Other: The Pelvic Proprioceptive Neuromuscular Facilitation Techniques Training
- Control Group (Active Comparator): The control group will receive patient education consisting of basic lumbar stabilization exercises 3 days a week for 6-weeks.
  Interventions: Other: The Patient Education

INTERVENTIONS:
Other: The Patient Education — The patient education will be given through a brochure and the content of the education included an exercise training consisting of simple exercises for lumbar stabilization (supine bridge, cat-camel, and lumbar stretching) and the participants will be asked to perform these exercises in 3 sets of 10 repetitions 3 days a week for 6-weeks.
Other: The Pelvic Proprioceptive Neuromuscular Facilitation Techniques Training — The content of the pelvic proprioceptive neuromuscular facilitation techniques training will include the application of the anterior depression pattern with the rhythmic initiation technique and the application of the posterior elevation pattern with the contract-relax stretch technique. All PNF techniques will be performed in 3 sets of 10 to 12 repetitions. The pelvic proprioceptive neuromuscular facilitation techniques training will be delivered face to face 3 days a week for 6 weeks by an experienced and trained physiotherapist.
  Arms: Experimental Group

SUMMARY:
The sacroiliac joint dysfunction (SIJD) which has a widely heterogeneous etiology, may cause impairment of stability, mobility, posture and flexibility as well as pain due to adaptive or pathological biomechanical changes. In 2020, the number of patients with low back pain (LBP) worldwide was more than half a billion and is expected to exceed 800 million by 2050. Although SIJD has been shown to be related with LBP in more than 30% of patients with LBP, SIJD is still often overlooked as a cause of LBP. Once the diagnosis of SIJD is confirmed by physical examination, the first treatment option consists of the use of a nonsteroidal anti-inflammatory drug or physiotherapy approaches. The proprioceptive neuromuscular facilitation (PNF) is a neurophysiological model-based multifaceted exercise method which is widely used in rehabilitation practice. However, despite the major role of SIJD among the causes of LBP, there are limited studies investigating the efficacy of PNF in SIJD and its effectiveness remains unclear. Thus, the aim of this study was to investigate the effect of pelvic PNF techniques on pain, mobility, flexibility, lumbar range of motion, posture, and trunk muscle endurance in patients with SIJD.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of SIJD
* Being between the ages of 18 and 40
* Volunteering to participate in the study

Exclusion Criteria:

* Having a history of any neurological, psychiatric and/or orthopedic disease
* Being pregnant or having a suspicion of pregnancy
* Having one or more of disc herniations, spondylosis, spondylolisthesis and/or similar lumbar pathologies that may cause low back pain
* Having a history of previous spine/hip/lower extremity surgery
* Having a history of active malignancy and/or infection
* Having a history of any injection and/or surgical procedure for the sacroiliac joint within the last 3 months

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
The Level of Low Back Pain | 6 weeks
  The intensity of low back pain will be rated subjectively on a 100-mm visual analog scale (VAS), where 0-mm indicated "no pain" and 100-mm indicated "worst possible pain"
Mobility | 6 weeks
  The Modified Schober's test will be used to assess mobility of lower back.
Flexibility | 6 weeks
  The sit-and-reach test will be used to assess flexibility of lower back.
Lumbar Range of Motion | 6 weeks
  A long-arm universal goniometer will be used to measure the lumbar range of motion. Flexion, extension, right and left lateral flexion, and right and left rotation will be assess.
Posture | 6 weeks
  The postural alignment will be assessed by using the New York Posture Rating Chart. Total score ranges between 13 and 65 points which higher scores indicate correct/normal postural alignment.
Trunk Muscle Endurance | 6 weeks
  Trunk flexor and extensor muscle endurance will be assessed with the flexor endurance test and Biering-Sørensen test, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Atlas University, Istanbul, Kagıthane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No